CLINICAL TRIAL: NCT04256954
Title: Peer Navigation for Individuals With Serious Mental Illness Leaving Jail
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Michigan State University (Other)
Collaborators: Brown University (Other)
Responsible Party: Principal Investigator, Maji Debena, Research Assistant Professor/ Principal Investigator, Michigan State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY00002543
Record Dates: First submitted 2020-01-06; First posted 2020-02-05 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Individuals With Serious Mental Illness Leaving Jails

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Peer navigation (Experimental): Those who are assigned to the intervention arm will receive peer navigation service by a trained peer navigator who will link them with mental health, medical and substance use services in the community.
  Interventions: Behavioral: Peer navigation intervention
- Standard of Care (No Intervention): SOC consists of TAU + monitoring and emergency referral, as is required to fulfil ethical obligations to trial participants. To determine the naturalistic effects and costs of adding peer navigation intervention, participants in both conditions can receive any other treatment available to them and we will not exclude participants receiving other treatment. We will carefully characterize TAU for each condition as part of our service utilization assessment.

INTERVENTIONS:
Behavioral: Peer navigation intervention — A peer navigator will assist those assigned to the intervention group access community mental health, medical care and substance use services. Peer navigators will help create linkages to services
  Arms: Peer navigation

SUMMARY:
Serious mental illness (SMI) is a burdensome and widely prevalent public health problem among incarcerated men and women. Incarcerated individuals with SMI re-entering the community after jail stay experience the double stigma of criminal justice involvement and having the diagnosis of SMI. As a result, they are likely to disengage with community level mental health, medical care and substance use services at re-entry. This study proposes the development and pilot test of peer navigator intervention to increase linkages to community level mental health, medical care and substance use services.

DETAILED DESCRIPTION:
Serious Mental Illness (SMI) is a stigmatized and disabling health condition that reduces average life expectancy by 25 years. SMI is also a prevalent public health problem affecting 25% of jail populations. Re-entry to the community following incarceration is a vulnerable time for justice-involved individuals with SMI, and SMI requires prompt and ongoing access to mental health and other healthcare services. Individuals with SMI who are re-entering the community following jail experience multiple barriers to access to community mental health, medical care (preventive and curative) and social services due to their debilitating symptoms, practical challenges accessing community services, and the stigma associated with being diagnosed with SMI. Peer navigation has been found to improve access to the mental health and medical care among individuals with SMI in the community. However, no peer support interventions for SMI have been tested to assist with mental health service linkage during re-entry to the community after incarceration. This study will develop and pilot test a peer navigator intervention for individuals with SMI re-entering the community after jail stay, providing formative work for a larger randomized controlled clinical trial evaluating the effectiveness of peer navigator intervention for justice-involved individuals with SMI. The intervention is based on social support theory. The project will: (a) develop a peer navigation intervention and evaluate its feasibility, acceptability, and potential engagement of target mechanisms for enrollment in mental health, medical care and substance use services among individuals with SMI re-entering the community after jail release and (b) conduct a randomized pilot trial in a sample of 40 individuals with SMI re-entering the community after jail release. Proposed target mechanisms include increased instrumental, informational, and emotional support for treatment engagement and recovery, as well as increased perception of social norms promoting treatment engagement and recovery. The control condition will be Standard Of Care (SOC). In addition to feasibility and acceptability, other outcomes include: (1) health service outcomes (primary) including enrollment/engagement/utilization of community mental health (primary), medical care and substance use services; and shorter days between release and first contact with healthcare provider; (2) Clinical outcomes: reduced psychiatric symptoms, increased functioning, adherence to psychiatric medications, fewer substance using days, fewer hospitalizations and suicide attempts; (3) Life context outcomes: nights unstably housed, and time until rearrest and (4) Potential target mechanisms that include instrumental, informational, and emotional support for treatment engagement and social norms about treatment engagement and recovery. Addressing the needs of re-entering individuals with SMI is a pressing priority for both the mental health and criminal justice systems. Peer navigators could play a critical role in continuing recovery and successful reintegration, reducing the impact of criminal justice involvement and mental health challenges.

ELIGIBILITY:
Inclusion Criteria:

* Incarcerated in the Genesee County Jail,
* Aged 18 or above,
* Has a lifetime DSM-5 diagnosis of SMI (including primary psychotic disorder [schizophrenia, schizoaffective disorder, or delusional disorder], bipolar disorder, and/or a major depressive disorder with psychotic features) as assessed by the Structured Clinical Interview for DSM-5 (SCID-5) and
* Anticipating release in the following two months.

Exclusion Criteria:

* Expect to be sentenced to prison (i.e., expect to go directly to prison, not home, from the jail),
* Cannot provide the name and contact information of at least two locator persons and/or
* Do not have access to any telephone.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2022-01-20 (Actual); Primary Completion 2024-02-22 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Feasibility: Client Satisfaction | 6 months after release
  Client Satisfaction Questionnaire- 8: scores range from 8-32, higher scores indicating higher satisfaction
Feasibility: End of treatment | 6 months after release
  End of Treatment Questionnaire: this is a descriptive measure, positive experiences described meaning higher feasibility of the service
Acceptability: Client Satisfaction Questionnaire | 6 months after release
  Client Satisfaction Questionnaire- 8: scores range from 8-32, higher scores indicating higher satisfaction
Acceptability: End of treatment | 6 months after release
  End of Treatment Questionnaire this is a descriptive measure, positive experiences described meaning better acceptability of the treatment

SECONDARY OUTCOMES:
Service linkage outcomes | Baseline, 3 months and 6 months
  Number of visits to outpatient as assessed by Treatment History Interview
Service linkage outcomes | Baseline, 3 months and 6 months
  Number of visits to emergency department as assessed by Treatment History Interview (THI)
Clinical outcomes | Baseline, 3 months and 6 months
  Presence of psychiatric symptoms as assessed by Altman Self-Rating Mania Scale; sum of items 1-5, with a cut off score of 6 or higher indicating presence of manic or hypomanic condition.
Clinical outcomes | Baseline, 3 months and 6 months
  Severity of psychiatric symptoms as assessed by Altman Self-Rating Mania Scale; scores range from 0-20, with a cut off score of 6 or higher indicating severity of psychiatric symptoms.
Clinical outcomes | Baseline, 3 months and 6 months
  Depressive symptoms as assessed by Quick Inventory of Depressive Symptoms; 16 questions, scores range from 0-27, higher scores indicating severity of depressive symptoms.
Clinical outcomes | Baseline, 3 months and 6 months
  Adherence to psychotropic medications as assessed by Brief Adherence Rating Scale; more days missed indicating poor adherence.
Clinical outcomes | Baseline, 3 months and 6 months
  Functioning as assessed by the 12-item WHO-Disability Assessment Schedule; scores range from 0-48, higher scores indicating greater functional impairment.
Clinical outcomes | Baseline, 3 months and 6 months
  Number of hospitalizations as assessed by Treatment History Interview
Clinical outcomes | Baseline, 3 months and 6 months
  Number of suicide attempts as assessed by Columbia Suicide Severity Rating Scale; scores range from 2-25, higher number indicating more intense suicidal ideation.
Clinical outcomes | Baseline, 3 months and 6 months
  Substance use (alcohol) as assessed by the Alcohol Use Disorders Identification Test
Clinical outcomes | Baseline, 3 months and 6 months
  Substance use (drugs) as assessed and Drug Use Disorders Identification Test
Target mechanisms | baseline, three months and six months.
  Self Stigma of Mental Illness Short Form
Life context outcomes | Baseline, 3 months and 6 months
  Number of nights unstably housed as measured by using calendar-based interview.
Life context outcomes | Baseline, 3 months and 6 months
  Days until rearrest as measured by using calendar-based interview.

CONTACTS AND LOCATIONS:
Locations (1):
- Genesee County Jail, Flint, Michigan, United States

IPD SHARING:
Plan to Share IPD: No